CLINICAL TRIAL: NCT01951105
Title: Corticostriatal Plasticity in the Transition to Chronic Pain: Effect of L-dopa
Brief Title: Effect of L-dopa In Subacute Back Pain Population
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Apkar Apkarian, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU00081444; R01DE022746 (NIH)
Record Dates: First submitted 2013-09-17; First posted 2013-09-26 (Estimated); Results first posted 2019-09-25 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Sub-acute Back Pain
Keywords: Subacute; Back; Pain; Brain; MRI
MeSH Terms: conditions — Pain | interventions — Naproxen; carbidopa, levodopa drug combination; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Observation (No Intervention): Individuals identified as having a recovering phenotype (SBPp) will be assigned to the observational arm and will be asked to continue his/her normal regime and return for the week 12 and week 24 visits for follow-up.
- Carbidopa/Levodopa & Naproxen (Active Comparator): Individuals identified as having a persisting phenotype (SBPr) will be treated with Carbidopa/Levodopa on a flexible dose-titration designed intervention based on dose-response TID throughout the 12 week treatment period.
  Naproxen (250mg) capsules will be administered orally, one capsule TID, throughout the 12 week treatment period.
  Interventions: Drug: Naproxen; Drug: Carbidopa/Levodopa
- Placebo & Naproxen (Placebo Comparator): Individuals identified as having a persisting phenotype (SBPr) will be treated with placebo capsule plus 250mg naproxen tablet three times a day for 12 weeks.
  Interventions: Drug: Naproxen; Drug: Placebo

INTERVENTIONS:
Drug: Naproxen — Take one 250mg naproxen tablet three times a day for 12 weeks.
  Other Names: Aleve; Anaprox; Antalgin; Apranax; Feminax Ultra; Flanax; Inza; Midol Extended Relief; Nalgesin; Naposin; Naprelan; Naprogesic; Naprosyn; Narocin; Proxen; Soproxen; Synflex; Xenobid
  Arms: Carbidopa/Levodopa & Naproxen; Placebo & Naproxen
Drug: Carbidopa/Levodopa — 12.5mg/50mg Carbidopa/Levodopa, administered orally as capsules, will be titrated up to TID over one week and then continued at that level for 4 weeks. If at the end of this initial 4 week period the participant has "responded," the subject will be maintained on that dose for the duration of the treatment period (12 weeks total). If there has not been a response, the dose will be increased to 25mg/100mg Carbidopa/Levodopa TID for the following 4 weeks at which time the pain status will be re-evaluated. If a response has occurred, that dose will be maintained in a blinded manner for the following 4 weeks of treatment; if not, further dose-titration will occur to 50mg/200mg Carbidopa/Levodopa TID for the final 4 weeks. If a subject experiences an AE at higher doses, then the subject will be given the next lower dose that s/he was able to tolerate and then be maintained on that dose for the remainder of the 12 week dosing period.
  Other Names: Sinemet
  Arms: Carbidopa/Levodopa & Naproxen
Drug: Placebo — Take two placebo capsules three times a day for 12 weeks.
  Other Names: Sugar Pill
  Arms: Placebo & Naproxen

SUMMARY:
This study aims to determine if early treatment with Carbidopa/Levodopa and Naproxen in individuals with sub-acute back pain (SBP) is associated with changes in blocking transition to chronic back pain (CBP).

DETAILED DESCRIPTION:
The transition from acute low back pain to chronic low back pain has been shown to be a result of changes in brain circuitry. Learning mechanisms give rise to the transition from acute to chronic pain and render the pain to become more emotional. The aim of this study is to further explore the idea that persistent pain, following an inciting injury, leads to an aversive learning signal that reorganizes the brain into a chronic pain state. We hypothesize that blocking the emotional/motivational learning response triggered by peripheral nerve injury in a critical time window will decrease the probability of transition to chronic pain. The primary hypothesis to be tested in the study is that early treatment with Carbidopa/Levodopa and Naproxen in individuals with sub-acute back pain (SBP) should decrease related reorganization and block transition to chronic back pain (CBP). This will be done through a 6 month, double-blind, randomized, placebo-controlled, three-arm, parallel-group trial of the pharmacological treatment Carbidopa/Levodopa for individuals (N = 200) with sub-acute back pain (SBP). A baseline MRI scan will be used to determine each subject's pain type and group assignment. Individuals with recovering sub-acute back pain will be observed over 6 months. Individuals with a persisting sub-acute back pain will be randomized to receive either 12 weeks of Carbidopa/Levodopa plus naproxen or placebo plus naproxen. The main outcome measurements will be the results of MRI scans at the baseline and final visit, assessment of back pain by the NRS pain scale, as well as pain assessment through self-reported questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, over the age of 18 years, (no racial/ethnic restrictions)
* Must have a history of low back pain for a minimum of 4 weeks and a maximum of 12 weeks with signs and symptoms of radiculopathy: positive straight leg raising test with dermatomal radiation and/or myotomal weakness and/or reflex asymmetry; pain must radiate into buttock or below
* Must have a high risk phenotype for chronification of back pain (evaluated at baseline T1-MRI, DTI-MRI, and fMRI scans)
* Must have an average pain score over a 5 day period (average of ~15 measures on smartphone app) immediately preceding the baseline visit of ≥ 5 (on a 0-10 NRS) at the baseline visit
* Must be willing to read and able to understand instructions as well as PROs
* Must be in generally stable health Must sign an informed consent document after complete explanation of the study documenting that they understand the purpose of the study, procedures to be undertaken, possible benefits, potential risks, and are willing to participate

Exclusion Criteria:

* Previous (distinct) episodes of back pain onset (more than 3 distinct episodes of back pain lasting for a total of more than 4 weeks) in the previous year
* Evidence of rheumatoid arthritis, ankylosing spondylitis, acute vertebral fractures, chronic spinal stenosis, prior back surgery and history of tumor of the spine
* Low back pain associated with any systemic signs or symptoms, e.g., fever, chills
* Other comorbid chronic pain conditions such as fibromyalgia or neuropathic pain secondary to diabetes or post-herpes zoster
* Chronic neurologic conditions, including Parkinson's disease, Alzheimer's disease, and other conditions associated with dementia
* Significant other medical disease such as congestive heart failure, coronary or peripheral vascular disease, chronic obstructive lung disease, or malignancy
* Diabetes Type I or Type II
* History of glaucoma or narrow angle glaucoma
* Presence of undiagnosed skin lesions or history of melanoma
* Presence of severe cardiovascular or pulmonary disease, bronchial asthma, renal, hepatic or endocrine disease
* History of myocardial infarction with residual cardiac arrhythmia
* History of gastrointestinal bleeding or peptic ulcer
* Diagnosis of current depression (assessed via BDI, total > 28 are excluded) or psychiatric disorder requiring treatment, or such a diagnosis in the previous 6 months
* Use of therapeutic doses of antidepressant medications (i.e., tricyclic antidepressants, SSRIs, SNRIs; low doses used only in the evening for sleep will be allowed if dose is not changed)
* Current use of recreational drugs or recent history of alcohol abuse (pattern of drinking having social, financial or physical consequences) or drug abuse
* Any change in medication for back pain in the last 30 days
* High dose opioid prophylaxis, defined as > 50mg morphine equivalent/day
* Use of MAOIs, currently or within the past 2 weeks
* Prior use of Levodopa
* Use of any of the following drugs: bromocryptine, linezolid, metoclopramide, phenothiazines,promethazine/codeine, isoniazid, rifampin, pyrazinamide
* Oral iron supplementation
* Contraindications to use of study product, based on any of the following:

  * Hypersensitivity to Carbidopa/Levodopa or other constituents of the Carbidopa/Levodopa capsules
  * Hypersensitivity to lactose or other constituents of the placebo capsules
  * Hypersensitivity to Naproxen or other constituents of the Naproxen capsules
  * Hypersensitivity to Acetaminophen or other constituents of the Acetaminophen tablets
* Currently taking Levodopa or dopaminergic drugs
* Involvement in litigation regarding their back pain or having a disability claim or receiving workman's compensation or seeking either as a result of their low back pain
* In the judgment of the investigator, unable or unwilling to follow protocol and instructions
* Intra-axial implants (e.g. spinal cord stimulators or pumps)
* All exclusion criteria for MR safety: any metallic implants, pacemaker, brain or skull abnormalities, tattoos on large body parts, and claustrophobia
* Pregnancy or inability to use an effective method of birth control in sexually active men and women while taking the study drug and for one week thereafter. Barrier contraceptives (condoms or diaphragm) with spermicide, intrauterine devices (IUD's), hormonal contraceptives, oral contraceptive pills, surgical sterilization, and complete abstinence are examples of effective methods of contraception.
* Following laboratory abnormalities: liver function tests (SGOT/SGPT) greater than twice the upper limit of normal; unexplained anemia (Hgb <9 g/dL); evidence of renal insufficiency (creatinine >upper limit of normal) or any other abnormality that the principal investigator feels puts the subject at risk during the study
* History of chronic opioid use for pain management.
* Any medical condition that in the investigator's judgment may prevent the individual from completing the study or put the individual at undue risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-02-24 (Actual); Primary Completion 2017-09-25 (Actual); Study Completion 2017-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Apkar Apkarian, PhD, Principal Investigator — Northwestern University Feinberg School of Medicine; Thomas J Schnitzer, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

REFERENCES:
- [Derived] Reckziegel D, Tetreault P, Ghantous M, Wakaizumi K, Petre B, Huang L, Jabakhanji R, Abdullah T, Vachon-Presseau E, Berger S, Baria A, Griffith JW, Baliki MN, Schnitzer TJ, Apkarian AV. Sex-Specific Pharmacotherapy for Back Pain: A Proof-of-Concept Randomized Trial. Pain Ther. 2021 Dec;10(2):1375-1400. doi: 10.1007/s40122-021-00297-2. Epub 2021 Aug 10. PMID 34374961

RESULTS

PARTICIPANT FLOW:
Groups:
- Observation: Individuals identified as having a recovering phenotype were assigned to the observational arm and were asked to continue his/her normal regime and return for the week 12 and week 24 visits for follow-up.
- Carbidopa/Levodopa & Naproxen: Individuals identified as having a persisting phenotype were randomized to oral Carbidopa/Levodopa on a flexible dose-titration designed intervention based on dose-response throughout the 12 week treatment period (12.5mg/50mg, 25mg/100mg, 50mg/200mg Carbidopa/Levodopa TID).
  Naproxen (250mg) capsules were administered orally, one capsule TID, throughout the 12 week treatment period.
- Placebo & Naproxen: Individuals identified as having a persisting phenotype were randomized to placebo capsule plus 250mg naproxen tablet TID for 12 weeks.
Period: Overall Study
Arm/Group | Observation | Carbidopa/Levodopa & Naproxen | Placebo & Naproxen
Started | 11 | 31 | 30
Completed 12 Weeks Treatment | 10 | 24 | 28
Completed | 10 | 21 | 28
Not Completed | 1 | 10 | 2
Not completed — Adverse Event | 0 | 5 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Observation | Carbidopa/Levodopa & Naproxen | Placebo & Naproxen | Total
Number analyzed (Participants) | 10 | 21 | 28 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data included in the analyses included all participants that completed the study
  years | 45.5 (12.0) | 49.1 (10.1) | 46.9 (13.2) | 47.5 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data included in the analyses included all participants that completed the study
  Participants
    Female | 3 | 7 | 14 | 24
    Male | 7 | 14 | 14 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data included in the analyses included all participants that completed the study
  Participants
    Hispanic or Latino | 2 | 1 | 6 | 9
    Not Hispanic or Latino | 8 | 19 | 20 | 47
    Unknown or Not Reported | 0 | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data included in the analyses included all participants that completed the study
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 2 | 8 | 10 | 20
    White | 7 | 12 | 17 | 36
    More than one race | 0 | 1 | 1 | 2
    Unknown or Not Reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 20% Reduction in Pain on the NRS Pain Intensity Scale
Description: Primary outcome is 20% reduction in pain intensity at p<0.1 based on pain ratings during 1 week prior to treatment and last week of study participation (at ~6months)
Time Frame: 6 months
Population: Note that one subject (out of 21) in the Carbidopa/Levodopa & Naproxen arm, and one subject (out of 28) in the Placebo & Naproxen arm, had missing NRS pain intensity scale ratings, hence they were excluded from primary outcome assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Observation | Carbidopa/Levodopa & Naproxen | Placebo & Naproxen
Number analyzed (Participants) | 10 | 20 | 27
Participants | 5 | 15 | 21
Statistical Analysis 1: Comparison: Carbidopa/Levodopa & Naproxen vs Placebo & Naproxen; Test type: Superiority; p = 1.0, Fisher Exact

2. Secondary Outcome: Percent of Residual Pain Stratified by Gender for Individuals Receiving Treatment
Description: Residual pain is computed based on pain ratings from the week prior to treatment and last week of study participation (at ~6months)
Time Frame: 6 months
Population: This outcome is limited to arms involving medication intake, thus it only concerns to Carbidopa/Levodopa & Naproxen (males and females) and Placebo & Naproxen (males and females). It does not include the observation arm. However numbers for the observation arm are also displayed.
Measure: Mean (Standard Error); unit: % residual pain
Groups:
- Carbidopa/Levodopa & Naproxen (Males): Male individuals identified as having a persisting phenotype were randomized to oral Carbidopa/Levodopa on a flexible dose-titration designed intervention based on dose-response throughout the 12 week treatment period (12.5mg/50mg, 25mg/100mg, 50mg/200mg Carbidopa/Levodopa TID).
  Naproxen (250mg) capsules were administered orally, one capsule TID, throughout the 12 week treatment period.
- Carbidopa/Levodopa & Naproxen (Females): Female individuals identified as having a persisting phenotype were randomized to oral Carbidopa/Levodopa on a flexible dose-titration designed intervention based on dose-response throughout the 12 week treatment period (12.5mg/50mg, 25mg/100mg, 50mg/200mg Carbidopa/Levodopa TID).
  Naproxen (250mg) capsules were administered orally, one capsule TID, throughout the 12 week treatment period.
- Placebo & Naproxen (Males): Male individuals identified as having a persisting phenotype were randomized to placebo capsule plus 250mg naproxen tablet TID for 12 weeks.
- Placebo & Naproxen (Females): Female individuals identified as having a persisting phenotype were randomized to placebo capsule plus 250mg naproxen tablet TID for 12 weeks.
- Observation (Males); Observation (Females): Individuals identified as having a recovering phenotype were assigned to the observational arm and were asked to continue his/her normal regime and return for the week 12 and week 24 visits for follow-up.
Arm/Group | Carbidopa/Levodopa & Naproxen (Males) | Carbidopa/Levodopa & Naproxen (Females) | Placebo & Naproxen (Males) | Placebo & Naproxen (Females) | Observation (Males) | Observation (Females)
Number analyzed (Participants) | 14 | 6 | 13 | 14 | 7 | 3
% residual pain | 62.97 (7.57) | 9.48 (3.12) | 37.96 (11.85) | 45.23 (9.86) | 85.55 (20.60) | 48.84 (30.27)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Observation | Carbidopa/Levodopa & Naproxen | Placebo & Naproxen
All-Cause Mortality (participants affected / at risk) | 0/11 | 1/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/11 | 3/31 | 0/30
Other Adverse Events (participants affected / at risk) | 0/11 | 17/31 | 14/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Observation (N=11) | Carbidopa/Levodopa & Naproxen (N=31) | Placebo & Naproxen (N=30)
Esophageal varices (Gastrointestinal disorders) | 0 | 1 | 0
Worsening angina (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Observation (N=11) | Carbidopa/Levodopa & Naproxen (N=31) | Placebo & Naproxen (N=30)
Upper Gastrointestinal (Gastrointestinal disorders) | 0 | 6 | 4
Headache (Nervous system disorders) | 0 | 3 | 3
Lower gastrointestinal (Gastrointestinal disorders) | 0 | 3 | 3
Drowsiness (General disorders) | 0 | 3 | 1
Lower respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Influenza (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-04-13): https://cdn.clinicaltrials.gov/large-docs/05/NCT01951105/Prot_SAP_000.pdf
  • Informed Consent Form (2017-04-13): https://cdn.clinicaltrials.gov/large-docs/05/NCT01951105/ICF_001.pdf